CLINICAL TRIAL: NCT06709456
Title: Drainage of Pleural Effusions in the Intensive Care Unit in Adults With Respiratory Failure: A Randomised Clinical Feasibility Trial of Performing Versus Withholding Pleural Drainage
Brief Title: Drainage Of Pleural Effusions in the Intensive Care Unit (DOPE-ICU) - Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olav Schjørring (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Olav Schjørring, Associate Professor, Consultant, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20240027; FID4401466 (Other Grant/Funding Number: Læge Sofus Carl Emil Friis og Hustru Olga Doris Friis' legat); 2024-0049 (Other Grant/Funding Number: Region Nordjyllands Sundhedsvidenskabelige Forskningsfond)
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Pleural Effusions; Respiratory Failure
Keywords: Pleural effusion; Respiratory failure; Pleural drainage; Ultrasonography; Intensive Care Unit; Randomised clinical trial; Feasibility; Critical care; Hypoxaemia; Hypercapnia
MeSH Terms: conditions — Pleural Effusion; Respiratory Insufficiency; Hypoxia; Hypercapnia

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, pragmatic, multicentre, open-label, randomised, parallel-group clinical feasibility trial
Masking Description: Blinding of statisticians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pleural drainage (Experimental): Ultrasonography-guided pleural drainage with insertion of a small-bore intrapleural catheter (typically pig-tail type catheter, size 6-14 French), conducted by e.g., intensivists or radiologists, as by local standards, of the pleural cavity with the estimated largest pleural effusion as soon as possible. A time interval of up to 24 hours from randomisation to intervention is expected. If bilateral pleural effusions ≥ 2 cm are present at randomisation, drainage of contralateral pleura should be conducted as soon as possible according to local standards, at least within 24 hours from insertion of the first pleural catheter unless pleural effusion has receded to < 2 cm prior to drainage. Inserted pleural catheters remain connected to a closed pleural drainage system, in situ and open until removed at clinicians' discretion according to local standards. New pleural effusion ≥ 2 cm during ICU stay within 90 days from randomisation will be drained similarly.
  Interventions: Procedure: Ultrasonography-guided pleural drainage
- No pleural drainage (No Intervention): No pleural drainage is conducted during ICU stay in 90 days from randomisation, unless escape protocol criteria are present being suspected or confirmed haemothorax, suspected or confirmed pneumothorax, suspected or confirmed pleural empyema, suspected or confirmed pleural malignancy, or indication for therapeutic pleural drainage as per the treating clinician and invasive or non-invasive mechanical ventilation or mask CPAP with arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) ratio ≤ 13.3 kPa in the most recent ABG analysis, high-flow humidified oxygen therapy with a flow ≥ 50 L/min and a PaO2/FiO2 ratio ≤ 13.3 kPa in the most recent ABG analysis, or persistent respiratory acidosis with a pH < 7.25 and an arterial partial pressure of carbon dioxide (PaCO2) > 6.0 kPa on the most recent ABG analysis in spite of non-invasive ventilation for > 1 hour.

INTERVENTIONS:
Procedure: Ultrasonography-guided pleural drainage — Ultrasonography-guided pleural drainage with insertion of a small-bore intrapleural catheter. Contralateral and repeated drainage conducted as specified during ICU stay until day 90.
  Arms: Pleural drainage

SUMMARY:
This trial evaluates the feasibility of ultrasound-guided pleural drainage versus no drainage in adult ICU patients with pleural effusions (fluid buildup around the lungs) and respiratory failure. Half of the patients will undergo drainage, while the other half will not unless their condition worsens to a prespecified degree. Outcomes include feasibility measures, clinical parameters, mortality, serious adverse events, and life support use over 90 days.

DETAILED DESCRIPTION:
Pleural effusions are common in intensive care unit (ICU) patients and are often treated with fluid drainage guided by ultrasonography. While this can improve oxygenantion levels, it is unclear whether it leads to better overall outcomes, and the procedure carries risks such as bleeding or lung collapse. There is limited evidence and no randomised trials supporting this procedure in ICU patients with respiratory failure. The DOPE-ICU feasibility trial will assess the feasibility of evaluating pleural drainage in such patients. Eligible ICU patients will be randomly assigned to either receive drainage or no drainage unless their condition worsens to a prespecified degree. Feasibility outcomes include the proportion of patients receiving drainage, protocol adherence, and proportion of patients with consent withdrawal for follow-up. Clinical outcomes include death rates, serious adverse events, and life support use, all within 90 days. Process outcomes include oxygenation, pH and arterial carbon dioxide tension at prespecified time points. The trial aims to determine whether a larger, more definitive trial is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Acute admission to the ICU.
* Age ≥ 18 years.
* Pleural effusion ≥ 2 cm in either pleural cavity assessed by ultrasonography, computed tomography or magnetic resonance imaging (measured between the parietal and visceral pleura perpendicularly to the chest wall at the largest-separation point).
* Respiratory failure defined as one or more of the following: any oxygen supplementation in an open system, invasive or non-invasive mechanical ventilation (including non-intermittent mask CPAP), or most recent arterial blood gas analysis with arterial partial pressure of carbon dioxide (PaCO2) > 6.0 kPa and pH < 7.35.

Exclusion Criteria:

* Mediastinal drain or pleural drain in situ on either side.
* Suspected or confirmed haemothorax (e.g., due to recent thoracic trauma or intrathoracic surgery).
* Suspected or confirmed pneumothorax (e.g., by anamnesis, on radiographic or ultrasonographic assessment, or by clinical presentation, e.g., due to presence of subcutaneous emphysema).
* Suspected or confirmed pleural empyema (e.g., by anamnesis or clinical presentation, or on CT, MRI or ultrasonographic assessment).
* Pleural malignancy (suspected or confirmed pleural lymphoma, pleural metastases or direct pleural invasion, or malignant mesothelioma).
* Antithrombotic treatment or coagulation deficiency incompatible with conducting pleural drainage as by local recommendations, and contraindications to reversal of this (clinical assessment).
* Clinically assessed absolute indication for therapeutic pleural drainage and:

  * invasive or non-invasive mechanical ventilation or mask CPAP with PaO2/FiO2 ratio ≤ 13.3 kPa in the most recent ABG analysis.
  * high-flow humidified oxygen therapy with a flow ≥ 50 L/min and a PaO2/FiO2 ratio ≤ 13.3 kPa in the most recent ABG analysis.
  * persistent respiratory acidosis with a pH < 7.25 and a PaCO2 > 6.0 kPa in the most recent ABG analysis in spite of non-invasive ventilation for > 1 hour.
* Withdrawal from active therapy or brain death deemed imminent.
* Expected ICU stay < 24 hours from randomisation.
* Pregnancy (in females < 60 years of age, non-pregnancy must be confirmed by a negative urine or plasma human chorionic gonadotropin, or presence a condition incompatible with pregnancy, e.g., previous hysterectomy, or conducted caesarean section during current hospitalisation).
* Under coercive measures (i.e., ongoing involuntary hospital admission or under correctional authorities' jurisdiction).
* Consent not obtainable as per Danish legislation.
* Previously randomised in the DOPE-ICU feasibility trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Intervention group separation (feasibility) | 90 days
  Proportion of patients receiving pleural drainage during ICU stay

SECONDARY OUTCOMES:
Protocol adhearence (feasibility) | 90 days
  Proportion of patients with one or more protocol violations defined as:
  * Participants allocated to pleural drainage who do not receive this within 24 hours from randomisation.
  * Participants allocated to pleural drainage with bilateral pleural effusion who do not receive the second (contralateral) pleural drainage within 24 hours from the primary drainage, unless pleural effusion has receded < 2 cm.
  * Participants allocated to no pleural drainage who receive pleural drainage at any time during ICU stay within 90 days from randomisation, including ICU readmissions, except when escape criteria for pleural drainage are present as specified (se "No intervention" arm).
Recruitment proportion (feasibility) | Through trial completion, estimated at 1 year.
  Proportion of included patients out of the number of eligible patients, i.e., patients who comply with all inclusion and exclusion criteria
Loss to follow-up (feasibility) | 90 days
  Proportion of participants without consent to the use of data
All-cause mortality (clinical outcome) | 90 days
  All-cause mortality
Serious adverse events (clinical outcome) | 90 days
  Proportion of patients with one or more serious adverse events (SAEs); SAEs are defined as new pneumothorax requiring invasive treatment (drainage or surgery), new haemothorax requiring red blood cell transfusion, new blood stream infection defined as any cultured microorganism from any blood sample except microorganisms clearly specified to be contaminants or likely contaminants by the microbiological department, and new episode of invasive mechanical ventilation defined as endotracheal intubation or re-intubation after extubation or tracheal decannulation.
Days alive without life support (clinical outcome) | 90 days
  Absolute number of days alive without life support being the use of mechanical ventilation, renal replacement therapy, or circulatory support
Days alive and out of hospital (clinical outcome) | 90 days
  Absolute number of days alive and out of hospital
Pleural infections (process outcome) | After 24 hours and within 90 days from randomisation
  Proportion of patients with new pleural infection after 24 hours from randomisation defined as any positive pleural fluid culture of any fungi or bacteria in any pleural fluid sampling conducted, except coagulase-negative Staphylococci, Enterococci, and Corynebacterium species, which will be considered contaminants.
24-hour oxygenation (process outcome) | 24 hours
  PaO2/FiO2 ratio in the arterial blood gas analysis conducted in ICU closest to 24 hours after randomisation.
72-hour oxygenation (process outcome) | 72 hours
  PaO2/FiO2 ratio in the arterial blood gas analysis conducted in ICU closest to 72 hours after randomisation.
24-hour pH (process outcome) | 24 hours
  pH in the arterial blood gas analysis conducted in ICU closest to 24 hours after randomisation.
72-hour pH (process outcome) | 72 hours
  pH in the arterial blood gas analysis conducted in ICU closest to 72 hours after randomisation.
24-hour carbon dioxide (process outcome) | 24 hours
  PaCO2 in the arterial blood gas analysis conducted in ICU closest to 24 hours after randomisation.
72-hour carbon dioxide (process outcome) | 72 hours
  PaCO2 in the arterial blood gas analysis conducted in ICU closest to 72 hours after randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Olav L Schjørring, MD, PhD, Principal Investigator — Department of Anaesthesia and Intensive Care, Aalborg University Hospital, Denmark
Locations (6):
- Denmark (6):
  - Department of Anaesthesia and Intensive Care, Aalborg University Hospital, Aalborg
  - ICU department 4131, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Anaesthesia and Intensive Care, Nordsjællands Hospital, University of Copenhagen, Hillerød, Hillerød
  - Department of Anaesthesiology and Intensive Care Medicine, Sygehus Lillebælt, Kolding, Kolding
  - Department of Anaesthesia and Intensive Care, Zealand University Hospital, Køge, Køge
  - Department of Anaesthesia and Intensive Care, Zealand University Hospital, Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
All original records (incl. consent forms, eCRFs, and relevant correspondences) will be archived at trial sites for 15 years. Anonymised data can be shared after primary publication upon specific request to the DOPE-ICU feasibility trial Steering Committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol with statistical analysis plan and informed consent forms are available on the webpage (www.cric.nu/dope-icu)
Access Criteria: Managed by the Steering Committee of the DOPE-ICU feasibility trial.

REFERENCES:
- See also: Related Info — http://www.cric.nu/dope-icu